CLINICAL TRIAL: NCT05001178
Title: Skeletal Maturation Within Different Skeletal Growth Patterns Using Cervical Vertebrae Maturation Index in Males.
Brief Title: Maturation Within Different Skeletal Growth Patterns Using Maturation Index in Males.
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Yehia Abdelghaffar Moustafa Saeda, Orthodontist Specialist, Cairo University
Other Study IDs: 12-5-21
Record Dates: First submitted 2021-08-04; First posted 2021-08-11 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-08

CONDITIONS: Skeletal Maturation
Keywords: cervical vertebrae maturation index

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (9):
- Class I horizontal grower
- Class I normal grower
- Class I vertical grower
- Class II horizontal grower
- Class II normal grower
- Class II vertical grower
- Class III horizontal grower
- Class III normal grower
- Class III vertical grower

SUMMARY:
The purpose of the study is to evaluate the difference between the maturation stages between different skeletal growth patterns

DETAILED DESCRIPTION:
comparing the maturation of different vertical and horizontal growth patterns using CVMI

ELIGIBILITY:
Inclusion Criteria:

* Only male patients between 8-16 years old with clear sharp cephalometric radiograph, the radiographs which have all the cervical vertebrae will be included in this study.

Exclusion Criteria:

* Previous orthodontic treatment.

  * Radiographs of poor quality.
  * Any hereditary diseases or syndromes such as Down's syndrome or cleidocranial dysostosis.
  * Any disease, trauma or fracture of the jaw that might have affected the normal growth of permanent dentition.

Ages: 8 Years to 16 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Study Population: males patients from 8 - 16 years
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2021-08 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
To evaluate the difference between the maturation stages (measured by CVMI index on lateral cephalograms) between different skeletal growth patterns | 8-16 years
  To evaluate the difference between the maturation stages (measured by CVMI index on lateral cephalograms) between different skeletal growth patterns

SECONDARY OUTCOMES:
to detect whether there were differences in the onsets of the pre-pubertal, pubertal and post-pubertal stages between the various antero-posterior and vertical skeletal patterns | 8-16 years
  to detect whether there were differences in the onsets of the pre-pubertal, pubertal and post-pubertal stages between the various antero-posterior and vertical skeletal patterns

CONTACTS AND LOCATIONS:
Overall Officials: Amr Eldakrory, Professor, Principal Investigator — Cairo University
Locations (1):
- Faculty of dentistry - Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mellion ZJ, Behrents RG, Johnston LE Jr. The pattern of facial skeletal growth and its relationship to various common indexes of maturation. Am J Orthod Dentofacial Orthop. 2013 Jun;143(6):845-54. doi: 10.1016/j.ajodo.2013.01.019. PMID 23726335
- [Background] Marceau K, Ram N, Houts RM, Grimm KJ, Susman EJ. Individual differences in boys' and girls' timing and tempo of puberty: modeling development with nonlinear growth models. Dev Psychol. 2011 Sep;47(5):1389-1409. doi: 10.1037/a0023838. PMID 21639623
- [Background] Cole TJ, Rousham EK, Hawley NL, Cameron N, Norris SA, Pettifor JM. Ethnic and sex differences in skeletal maturation among the Birth to Twenty cohort in South Africa. Arch Dis Child. 2015 Feb;100(2):138-43. doi: 10.1136/archdischild-2014-306399. Epub 2014 Nov 19. PMID 25409981
- [Background] Soegiharto BM, Moles DR, Cunningham SJ. Discriminatory ability of the skeletal maturation index and the cervical vertebrae maturation index in detecting peak pubertal growth in Indonesian and white subjects with receiver operating characteristics analysis. Am J Orthod Dentofacial Orthop. 2008 Aug;134(2):227-37. doi: 10.1016/j.ajodo.2006.09.062. PMID 18675204
- [Background] Kim JH, Viana MA, Graber TM, Omerza FF, BeGole EA. The effectiveness of protraction face mask therapy: a meta-analysis. Am J Orthod Dentofacial Orthop. 1999 Jun;115(6):675-85. doi: 10.1016/s0889-5406(99)70294-5. PMID 10358251
- [Background] Nanda SK. Patterns of vertical growth in the face. Am J Orthod Dentofacial Orthop. 1988 Feb;93(2):103-16. doi: 10.1016/0889-5406(88)90287-9. PMID 3422525
- [Background] Kuc-Michalska M, Baccetti T. Duration of the pubertal peak in skeletal Class I and Class III subjects. Angle Orthod. 2010 Jan;80(1):54-7. doi: 10.2319/020309-69.1. PMID 19852640
- [Background] Jeelani W, Fida M, Shaikh A. The duration of pubertal growth peak among three skeletal classes. Dental Press J Orthod. 2016 Sep-Oct;21(5):67-74. doi: 10.1590/2177-6709.21.5.067-074.oar. PMID 27901231
- [Background] Baccetti T, Franchi L, McNamara JA Jr. An improved version of the cervical vertebral maturation (CVM) method for the assessment of mandibular growth. Angle Orthod. 2002 Aug;72(4):316-23. doi: 10.1043/0003-3219(2002)0722.0.CO;2. PMID 12169031
- [Background] Buschang PH, Tanguay R, Demirjian A, LaPalme L, Turkewicz J. Mathematical models of longitudinal mandibular growth for children with normal and untreated Class II, division 1 malocclusion. Eur J Orthod. 1988 Aug;10(3):227-34. doi: 10.1093/ejo/10.3.227. No abstract available. PMID 3181302